CLINICAL TRIAL: NCT05862896
Title: Exploring Gas Transfer and the Utility of Dynamic Chest Radiography in Long Covid Patients.
Acronym: LoCTDC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: LHS0056
Record Dates: First submitted 2023-05-16; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy, age and sex matched controls
- Long Covid: Patients with breathlessness (defined as self-reported modified Borg Scale score of 2 or more when walking on flat ground for 100 metres) that has continued or developed and persists more than 4 weeks after acute COVID 19 i.e., related to 'long COVID' (covid confirmed by photographic evidence of positive lateral flow/NHS application, EMIS records or hospital lab data).

SUMMARY:
This study aims to identify if breathless patients with Long COVID have reduced transfer factor on pulmonary function testing and if the degree of transfer factor reduction is correlated with the symptom severity and physiological ability to exercise. We will also investigate whether a new type of X-ray called a dynamic chest X-ray can identify perfusion abnormalities and whether these correlate with differences in diffusion capacity measured on a pulmonary function test.

DETAILED DESCRIPTION:
Long COVID is the term used to describe patients who present with persistent symptoms after recovering from SARS-CoV-2 infection. Patients exhibit a range of symptoms and commonly report respiratory and cardiac phenomena including breathlessness, feeling tight chested and having persistent tachycardias. Survey data suggests up to 87% of patients discharged from hospital after COVID-19 infection have ongoing symptoms 60 days after discharge, with 43% describing breathlessness. In the USA, 35% of patients treated for SARS-CoV-2 as an outpatient have ongoing symptoms, with a similar percentage of the population unable to return to their normal work. The natural history and pathophysiology of long COVID is not yet fully understood. Few studies have explored pulmonary function in post-COVID patients. There are suggestions that functional limitation is related to lung abnormalities affecting both ventilation (air flow) and perfusion (blood flow), possibly caused by micro-blood clots. Establishing a relatively cost-effective and accessible way of diagnosing these will allow clinicians to treat or signpost the patients to the correct services. This is vital at both the patient and health system level.

Full pulmonary function testing is routinely done in respiratory clinics to investigate breathlessness and diagnose conditions such as asthma, chronic obstructive pulmonary disease (COPD) and pulmonary fibrosis. It includes a measure of transfer factor, an estimate of the efficiency of the diffusion of gas from the lung into the blood stream. The lungs' ability to absorb carbon monoxide (CO) is measured as a proxy for the ability to absorb oxygen. It is hypothesised that long COVID patients with breathlessness have abnormal gas transfer due to lung tissue damage at an alveolar level and/or perfusion abnormalities such as micro clots. Dynamic X-ray is a new, innovative technology to image the thoracic cavity throughout the breathing cycle allowing assessment of pulmonary function and possibly diagnose small ventilation-perfusion abnormities. Liverpool hosts the only dynamic X-ray machine in Europe. Potential applications beyond COVID are numerous, including filling diagnostic gaps in many lung diseases where expensive lung function testing is an unrealistic possibility in the medium term.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (over 18 years old)
2. Patients with breathlessness (defined as self-reported modified Borg Scale score of 2 or more when walking on flat ground for 100 metres) that has continued or developed and persists more than 4 weeks after acute COVID 19 i.e., related to 'long COVID' (covid confirmed by photographic evidence of positive lateral flow/NHS application, EMIS records or hospital lab data).
3. Able to achieve positioning for a PA chest X-ray for a 20 second period
4. Able to hold their breath for at least 7 seconds
5. Fluent spoken English - to ensure a comprehensive understanding of the research project and their proposed involvement
6. Able to provide written informed consent
7. For control group: Age, sex matched to participants identified in the affected group

Exclusion Criteria:

1. Any contraindication to pulmonary function testing or DCR
2. Pregnancy
3. For women of childbearing age, a positive pregnancy test or refusal of pregnancy test (a negative urinary pregnancy test on the day of DCR is a requirement)
4. Significant other respiratory co-morbidities as judged by study clinician
5. Significant research related radiation exposure in last 12 months prior to consent (from participation in a previous studies involving radiation exposure, with a research dose constraint of 0.4 mSv)
6. Unable to provide informed consent for any reason
7. For the long covid arm no evidence of a positive covid-19 test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of adults (over 18 years) with breathlessness secondary to long COVID identified in the community will be compared with a control group of age and sex matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 12 months
  1) To establish the proportion of patients with long COVID that have abnormal transfer factor on pulmonary function testing.